CLINICAL TRIAL: NCT01271621
Title: Influence of Glidescope Assisted Endotracheal Intubation on Intraocular Presure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RP 1013
Record Dates: First submitted 2010-11-15; First posted 2011-01-07 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Effect of Intubation on Intraocular Pressure
Keywords: Airtraq, Intraocular pressure
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macintoch group (Active Comparator): Intubation with Macintoch Laryngoscope
  Interventions: Device: Intubation
- Glidescope (Experimental): Inubation by Glidescope
  Interventions: Device: Intubation

INTERVENTIONS:
Device: Intubation — Endotracheal intubation

SUMMARY:
Tracheal intubation with traditional Macintosh laryngoscope is associated with increase in intraocular pressure along with tachycardia and hypertension. These effects are not desirable in ophthalmic patients especially in patients with glaucoma. GlideScope video laryngoscope system is a new approach for laryngoscopy and tracheal intubation. It does not require a direct line of sight to the glottis when intubating with the Glidescope and as a result intubation is much less stimulating to the patient. Therefore GlideScope video laryngoscope assisted intubation could be a preferable technique for intraocular surgery offering advantages in terms of intraocular pressure and cardiovascular stability.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2 with normal intra-ocular pressure.

Exclusion Criteria:

* history or occurrence of difficult intubation.
* presence of previous anterior segment pathology.
* previous intraocular surgery.
* patients with history of glaucoma.
* brain pathology and other neurological disorder which might affect to their intraocular pressure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | one year

CONTACTS AND LOCATIONS:
Locations (1):
- king Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia